CLINICAL TRIAL: NCT04323488
Title: Neural Mechanisms of Successful Intervention in Children With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jason Yeatman, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 52231; R01HD095861-01A1 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Dyslexia, Developmental
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: subjects are seen before and after receiving 8 weeks of reading instruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lindamood-Bell Seeing Stars (Experimental): Subjects receive reading instruction focusing on the building blocks of reading
  Interventions: Behavioral: Lindamood-Bell Seeing Stars
- Control (No Intervention): Subjects are followed longitudinally but do not receive intervention

INTERVENTIONS:
Behavioral: Lindamood-Bell Seeing Stars — Seeing Stars in a curriculum developed by Lindamood-Bell. It is published and openly available. It involves systematic training in the building blocks of skilled reading.
  Arms: Lindamood-Bell Seeing Stars

SUMMARY:
Dyslexia, an impairment in accurate or fluent word recognition, is the most common learning disability affecting roughly ten percent of children. This proposal capitalizes on cutting edge neuroimaging methods, in combination with reading education programs, to generate a new understanding of how successful reading education shapes the development of the brain circuits that support skilled reading. A deeper understanding of the mechanisms of successful remediation of dyslexia, and individual differences in learning, will pave the way for personalized approaches to dyslexia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Reading difficulties defined as low scores on standardized measures of reading skills

Exclusion Criteria:

* no major contraindication for MRI (braces, metal implants, pacemakers, vascular stents, or metallic ear tubes).
* Because the study involves measurements of reading and language ability, new recruits will be native English speakers.
* Subjects have no history of neurological disorder, significant psychiatric problems
* exclude claustrophobic subjects since an MRI might be uncomfortable for them.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Yeatman, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
All consent forms in the Yeatman lab contain a data sharing clause that allows de-identified data to be shared publicly. The lab policy is that data and analysis code are always publicly released to accompany each published manuscript from the lab. This policy ensures that published findings can be reproduced by other researchers and the general public. In our experience, this also creates a useful resource to document our methods, describe methodological decisions in greater detail than afforded by journal articles, and publicly release datasets that may be of utility to other researchers. Data and code are organized into a well-documented repository (see https://github.com/yeatmanlab) with a persistent digital identifier ensuring that it will be available in perpetuity. Within the repository is documentation to reproduce each manuscript figure and each reported statistic. The lab is a strong proponent of open science and has adhered to this lab policy for every published manuscript.

REFERENCES:
- [Result] Stone HL, Mitchell JL, Fuentes-Jimenez M, Tran JE, Yeatman JD, Yablonski M. Anatomically distinct regions in the inferior frontal cortex are modulated by task and reading skill. J Neurosci. 2025 Mar 24;45(19):e1767242025. doi: 10.1523/JNEUROSCI.1767-24.2025. Online ahead of print. PMID 40127940

RESULTS

PARTICIPANT FLOW:
Groups:
- Lindamood-Bell Seeing Stars: Subjects receive reading instruction Lindamood-Bell Seeing Stars that focuses on systematic training in the building blocks of skilled reading.
Period: Overall Study
Arm/Group | Lindamood-Bell Seeing Stars | Control
Started | 44 | 46
Began study procedures | 44 | 43
Completed | 40 | 37
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lindamood-Bell Seeing Stars | Control | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 46 | 90
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 23 | 24 | 47
  Non-binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 28 | 24 | 52
  More than one race | 2 | 4 | 6
  Other | 4 | 4 | 8
  Prefer not to answer | 1 | 0 | 1
  Not reported/unknown | 0 | 5 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: White Matter Plasticity - Left Arcuate Tract
Description: Change in white matter mean diffusivity (MD) measured with diffusion MRI. MD quantifies the average magnitude of water diffusion within a given region of tissue. An increase in mean diffusivity (MD) suggests an increase in free water movement (corresponds to less white matter integrity), while a decrease in MD suggests restricted water diffusion, potentially from increased cellular density (corresponds to greater white matter integrity). Values typically range from approximately 0.5 to 1.5 × 10^-3 mm²/s in healthy white matter.
Time Frame: Baseline (within 2 weeks pre-intervention), post-intervention (within 2 weeks post-intervention, up to 10 weeks), and at 1 year follow up
Population: Participants with readable scans (i.e., low-movement, high quality) at the respective time point
Measure: Mean (Standard Deviation); unit: mm^2/s
Arm/Group | Lindamood-Bell Seeing Stars | Control
Number analyzed (Participants) | 44 | 37
mm^2/s
  baseline: number analyzed (Participants) | 44 | 33
  baseline | 0.837 (0.039) | 0.838 (0.033)
  2 weeks post-intervention: number analyzed (Participants) | 26 | 37
  2 weeks post-intervention | 0.842 (0.041) | 0.844 (0.038)
  1 year follow-up: number analyzed (Participants) | 39 | 23
  1 year follow-up | 0.839 (0.038) | 0.830 (0.038)
Statistical Analysis 1: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.925, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Control; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.834, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.180, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: Control; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.091, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

2. Primary Outcome: White Matter Plasticity - Inferior Longitudinal Tract
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants with readable scans (i.e., low-movement, high quality) at the respective time point
Measure: Mean (Standard Deviation); unit: mm^2/s
Arm/Group | Lindamood-Bell Seeing Stars | Control
Number analyzed (Participants) | 44 | 37
mm^2/s
  baseline: number analyzed (Participants) | 44 | 33
  baseline | 0.963 (0.036) | 0.957 (0.028)
  2 weeks post-intervention: number analyzed (Participants) | 26 | 37
  2 weeks post-intervention | 0.963 (0.034) | 0.956 (0.035)
  1 year follow-up: number analyzed (Participants) | 39 | 23
  1 year follow-up | 0.957 (0.040) | 0.952 (0.039)
Statistical Analysis 1: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.524, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Control; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.379, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.010, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: Control; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.017, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

3. Primary Outcome: Visual Word Form Area (VWFA) Size
Description: Visual Word Form Area (VWFA) refers to a region in the brain associated with the recognition of written words. VWFA size is calculated as the number of vertices in the cotrical surface. There are no definitive clinical relevant thresholds for the size of the VWFA that apply universally. Research indicates that variations in VWFA size and activation are associated with reading abilities and disorders.
Time Frame: as for outcome 1
Population: Participants with readable scans (i.e., low-movement, high quality) at the respective time point
Measure: Mean (Standard Deviation); unit: vertices
Arm/Group | Lindamood-Bell Seeing Stars | Control
Number analyzed (Participants) | 42 | 42
vertices
  baseline | 142.00 (178.71) | 302.74 (385.92)
  2 weeks post-intervention: number analyzed (Participants) | 29 | 40
  2 weeks post-intervention | 146.69 (179.47) | 282.40 (372.00)
  1 year follow-up: number analyzed (Participants) | 40 | 25
  1 year follow-up | 375.53 (363.50) | 337.20 (333.21)
Statistical Analysis 1: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.60, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Control; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.03, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.60, t-test, 2 sided
Statistical Analysis 4: Comparison: Control; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.03, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

4. Primary Outcome: Woodcock-Johnson Basic Reading Skills (WJ BRS) Assessment Battery
Description: The Woodcock-Johnson Basic Reading Skills (WJ BRS) Assessment Battery results in a composite score across multiple assessments. Assessment scores are transformed to create an overall score range of 0 to 200. A score of 100 indicates average reading ability. Scores below 85 may indicate potential reading difficulties
Time Frame: as for outcome 1
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lindamood-Bell Seeing Stars | Control
Number analyzed (Participants) | 44 | 43
score on a scale
  baseline | 80.75 (10.52) | 96.85 (17.30)
  2 weeks post-intervention: number analyzed (Participants) | 43 | 43
  2 weeks post-intervention | 88.33 (9.90) | 96.02 (19.20)
  1 year follow-up: number analyzed (Participants) | 40 | 29
  1 year follow-up | 89.95 (8.50) | 95.10 (16.97)
Statistical Analysis 1: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p < 0.001, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Control; Within-group analysis of change from baseline and post-intervention (within 2 weeks post-intervention); Test type: Other; p = 0.29, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Lindamood-Bell Seeing Stars; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p < 0.001, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: Control; Within-group analysis of change from baseline and 1 year follow up; Test type: Other; p = 0.26, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: Up to 2.5 years
Arm/Group | Lindamood-Bell Seeing Stars | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT04323488/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT04323488/ICF_001.pdf